CLINICAL TRIAL: NCT05644093
Title: Open-label, Cross-over Study of IM and IV Doses of SPL026 in Healthy, Psychedelic-experienced Participants (Part A: IM and IV Doses) and Participants With Little to no Psychedelic Experience (Part B: IM Dose Only)
Brief Title: IM and IV SPL026 Drug Product in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Small Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CT026_003
Record Dates: First submitted 2022-11-17; First posted 2022-12-09 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychedelic Experienced IM then IV crossover (Experimental): Participants will be dosed with IM SPL026 then IV SPL026 2-3 weeks later.
  Interventions: Drug: SPL026 IV; Drug: SPL026 IM
- Psychedelic Naive IM dosing only (Experimental): Participants will be dosed with IM SPL026 one time.
  Interventions: Drug: SPL026 IM

INTERVENTIONS:
Drug: SPL026 IV — IV dosing
  Other Names: DMT
  Arms: Psychedelic Experienced IM then IV crossover
Drug: SPL026 IM — IM dosing
  Other Names: DMT

SUMMARY:
The goal of this clinical trial is to test SPL026 given via injection into a muscle in healthy volunteers.

DETAILED DESCRIPTION:
Part A: Crossover IM then IV dosing with SPL026 in psychedelic experienced, healthy volunteers.

PART B: IM dosing only with SPL026 in less experienced/psychedelic naive, healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

Part A only

1. Healthy psychedelic-experienced female or male participants (psychedelic-experienced is defined as having at least 2 previous experiences, with breakthrough, of serotonergic psychedelic drugs, including but not limited to: DMT, ayahausca, LSD, LSA [morning glory seeds], DOI [2,5-Dimethoxy-4- iodoamphetamine], DOB [dimethoxybromoamphetamine], DOC [2,5- Dimethoxy-4-chloroamphetamine], 2CB [2-(4-bromo-2,5- dimethoxyphenyl)ethanamine], 2CE [1-(2,5-Dimethoxy-4-ethylphenyl)-2- aminoethane], mescaline, peyote, san pedro, ibogaine and psilocybin [including mushroom species containing psilocybin]).
2. No psychedelic drug use within 6 weeks prior to dosing.

   Part B only
3. Healthy female or male participants with little to no psychedelic experience (defined as having never taken serotonergic psychedelic drugs, or have only taken sub-breakthrough doses of serotonergic psychedelic drugs, in any form, < 5 times, including but not limited to: DMT, ayahuasca, LSD, LSA, DOI, DOB, DOC, 2CB, 2CE, mescaline, peyote, san pedro, ibogaine and psilocybin [including mushroom species containing psilocybin]).
4. No psychedelic drug use within 6 months prior to dosing.

   Parts A and B
5. Aged 25-65 years.
6. A body mass index (BMI; Quetelet index) in the range 18.0-33.9 kg/m2. Body Mass Index =
7. Sufficient intelligence to understand the nature of the trial and any hazards of participating in it. Ability to communicate satisfactorily with the investigator and to participate in, and comply with the requirements of, the entire trial.
8. Willingness to give written consent to participate after reading the information and consent form, and after having the opportunity to discuss the trial with the investigator or his delegate.
9. Agree to follow the contraception requirements of the trial.
10. Agree not to donate blood or blood products during the study and for up to 3 months after the (last) administration of the trial medication.
11. Willing to refrain from psychedelic drug use (excluding the study drug) during the trial and until the follow up call.
12. Willingness to give written consent to have data entered into The Overvolunteering Prevention System (TOPS).
13. Willing to be contacted by email and video call, and have online access.
14. Has veins deemed suitable for cannulation (IV infusion and/or blood sampling).

Exclusion Criteria:

1. Current or previously diagnosed mental health disorder as defined by Diagnostic and Statistical Manual of Mental Disorders (DSM-V) criteria.
2. First degree relative with schizophrenia spectrum or other psychotic disorders, or bipolar and related disorders.
3. Disposition judged by the investigator (or delegate) to be incompatible with establishment of rapport with therapy team and/or safe exposure to DMT.
4. Woman who is pregnant or lactating, or pre-menopausal woman who is sexually active and not using a reliable method of contraception (see section 11).
5. Clinically relevant abnormal history, physical findings, ECG, or laboratory values at the pre-trial screening assessment that could interfere with the objectives of the trial or the safety of the participant.
6. Presence of acute or chronic illness, condition or infection, or history of chronic illness or condition (including psychological and neurological [eg seizure] disorder) considered sufficient to invalidate the participant's participation in the trial or make it unnecessarily hazardous.
7. Impaired endocrine, thyroid, hepatic, respiratory or renal function, diabetes mellitus, coronary heart disease or any of the following cardiovascular conditions: arrhythmia, a clinically significant screening ECG abnormality or family history of long QT syndrome or sudden death, artificial heart valve, current or any history of hypertension, or any other significant current or history of cardiovascular condition, that may affect safety in the opinion of the investigator.
8. History of serious suicide attempts (ie those that require hospitalisation); as assessed by the BSS.
9. Presence or history of severe adverse reaction to any drug or a history of sensitivity to serotonergic psychedelic drugs.
10. Use of a prescription medicine (except oral contraceptives or any hormone therapy), certain herbal supplements (eg St John's Wort, to be reviewed by trial physician), or over-the-counter medicine, during the 28 days before the first dose of trial medication. Use of acetaminophen (paracetamol) and non-steroidal anti-inflammatory drugs (eg ibuprofen) are permitted up to 4 h before the first dose of trial medication.
11. Receipt of an investigational product (including prescription medicines) as part of another clinical trial within the 3 months before (first) admission to this study; in the follow-up period of another clinical trial at the time of screening for this study.
12. Presence or history of drug or alcohol abuse, or intake of more than 14 units of alcohol weekly.
13. Daily cannabis use or cannabis dependence as defined by ICD10.
14. Use of cannabis in the 24 h before each study visit.
15. Evidence of drug abuse on urine testing (with the exception of cannabis).
16. Unable to be nicotine free (refrain from smoking or nicotine-containing products) for 24 h before and until the morning after dosing.
17. Blood pressure and pulse rate in the supine and standing position at the screening examination outside the ranges: blood pressure 80-150 mm Hg systolic; 30-100 mm Hg diastolic; pulse rate 40-100 beats/min. Borderline values (ie values that are within 5 mm Hg of the range for blood pressure or 5 beats/min of the range for pulse rate) will be repeated. Participants can be included if the repeat value is within range or still borderline but deemed not clinically significant by the investigator.
18. QTcF value at screening greater than 450 msec (men) or 470 msec (women) on 12-lead ECG. Triplicate measurements will be made, and a mean QTcF value higher than 450 msec (men) or 470 msec (women) will lead to exclusion. A repeat (in triplicate) is allowed on one occasion for determination of eligibility.
19. Possibility that the participant will not cooperate with the requirements of the protocol.
20. Positive test for hepatitis B, hepatitis C or human immunodeficiency virus (HIV).
21. Loss of more than 400 mL blood during the 3 months before the trial, eg as a blood donor.
22. Phobia of needles or blood.
23. Objection by General Practitioner (GP) to participant entering trial.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2023-04-05 (Actual); Study Completion 2023-04-05 (Actual)

PRIMARY OUTCOMES:
Lab biochemistry [Safety & Tolerability] | Change from baseline at Day 1 post dose
  Values of potential clinical importance
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Throughout the study until 14 days after dosing (Day 15 EOS)
  Adverse Events (AEs)
Heart Rate [Vital Signs - Safety & Tolerability] | Change from baseline heart rate at Day 1 or Day 2 post dose
  pulse rate will be measured in bpm
Blood Pressure [Vital Signs - Safety & Tolerability] | Change from baseline blood pressure at Day 1 or Day 2 post dose
  arterial blood pressure
Temperature [Vital Signs - Safety & Tolerability] | Change from baseline temperature at Day 1 or Day 2 post dose
  tympanic temperature
12-lead ECG [Safety & Tolerability] | Change from baseline ECG at Day 1 or Day 2 post dose
  QTcX intervals
Physical Exam [Safety & Tolerability] | Change from baseline at Day 1 post dose
  Full physical exam screening and a brief symptom guided exam at Day -1 and Day 1
Beck Scale for Suicidal Ideation (BSS) - [Safety & Tolerability] | Change from baseline at Day 15 post dose
  The Beck Suicidal Ideation scale to monitor suicidal ideation

SECONDARY OUTCOMES:
Evaluation of plasma levels of DMT | Day 1
  Pharmacokinetic parameter calculation
Mystical Experience Questionnaire (MEQ) - [Pharmacodynamics - Psychometric Scales and Questionnaires] | Day 1 (dosing day)
  Compare MEQ between different routes of administration (IV & IM)
Challenging Experience Questionnaire (CEQ) - [Pharmacodynamics - Psychometric Scales and Questionnaires] | Day 1 (dosing day)
  Compare CEQ between different routes of administration (IV & IM)

CONTACTS AND LOCATIONS:
Overall Officials: Adeep Puri, MD, Principal Investigator — HMR
Locations (1):
- Hammersmith Medicines Research, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan for this yet.

REFERENCES:
- See also: Location of Clinical Study Report Synopsis — https://www.isrctn.com/ISRCTN63723571